CLINICAL TRIAL: NCT02134925
Title: Randomized, Double-Blind, Placebo-Controlled Trial of MUC1 Vaccine in Patients With Newly Diagnosed Advanced Adenomas
Brief Title: Vaccine Therapy in Treating Patients With Newly Diagnosed Advanced Colon Polyps
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2014-01080; NCI-2014-01080 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HHSN261201200042I; N01-CN-2012-00042; MAY2013-01-01 (Other: Mayo Clinic in Rochester); MAY2013-01-01 (Other: DCP); N01CN00042 (NIH); P30CA015083 (NIH); NCT02886000 (obsolete NCT alias)
Record Dates: First submitted 2014-05-07; First posted 2014-05-09 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Colorectal Adenoma; Colorectal Adenoma With Severe Dysplasia; Colorectal Carcinoma; Colorectal Tubulovillous Adenoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (MUC1 peptide-poly-ILCLC adjuvant vaccine) (Experimental): Participants receive MUC1 peptide-poly-ICLC adjuvant vaccine SC in weeks 0, 2 and 10 and a booster injection in week 53.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: MUC1 Peptide-Poly-ICLC Vaccine; Other: Quality-of-Life Assessment
- Arm II (saline) (Placebo Comparator): Participants receive saline SC in weeks 0, 2, and 10 and a booster injection in week 53.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Saline

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: MUC1 Peptide-Poly-ICLC Vaccine — Given SC
  Arms: Arm I (MUC1 peptide-poly-ILCLC adjuvant vaccine)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Saline — Given SC
  Other Names: ISOTONIC SODIUM CHLORIDE SOLUTION; Normal Saline; Sodium Chloride 0.9%
  Arms: Arm II (saline)

SUMMARY:
This randomized phase II clinical trial studies how well MUC1 peptide-poly-ICLC adjuvant vaccine works in treating patients with newly diagnosed advanced colon polyps (adenomatous polyps). Adenomatous polyps are growths in the colon that may develop into colorectal cancer over time. Vaccines made from peptides may help the body build an effective immune response to kill polyp cells. MUC1 peptide-poly-ICLC adjuvant vaccine may also prevent the recurrence of adenomatous polyps and may prevent the development of colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the immunogenicity at week 12 of a MUC1 peptide vaccine with adjuvant (MUC1 peptide-poly-ICLC adjuvant vaccine) (administered at 0, 2, and 10 weeks) in participants with a history of an advanced adenoma, randomized to receive MUC1 peptide vaccine versus placebo.

SECONDARY OBJECTIVES:

I. To evaluate the ability of the vaccine to elicit a long-term memory response.

II. To compare the adenoma recurrence rate from surveillance exams occurring at least 1 year and up to 3 years after week 0 vaccine administration - MUC1 versus placebo.

III. To compare the adenoma recurrence rates between MUC1 and placebo by excluding the following types of adenomas: participants with adenomas =< 5 mm; participants with adenomatous tissue which may represent residual adenoma at the site of the previous advanced adenoma; participants with adenomatous tissue detected in the same segment of the bowel as the previous advanced adenoma.

IV. To assess adverse events to the MUC1 peptide vaccine in comparison to placebo during Parts I and II.

V. To assess patient reported injection site reaction events from the Vaccine Report Card.

TERTIARY OBJECTIVES:

I. To compare the anti-MUC1 antibody titer at the time of surveillance colonoscopy for the purpose of evaluating the anti-MUC1 antibody response in relation to adenoma recurrence.

II. To evaluate MUC1 expression on baseline advanced adenomas and on recurrent adenomas detected at surveillance colonoscopy.

III. To evaluate levels of circulating myeloid derived suppressor cells (MDSC) in the vaccinated and the placebo group and correlate with anti-MUC1 antibody levels and adenoma recurrence.

IV. To establish a biospecimen repository archive including live cells, plasma, and germline deoxyribonucleic acid (DNA) for future immunologic (e.g. MUC1-specific T cells) and other assays (systems biology approach to detect differences between responders and non-responders), testing not currently accommodated within the budget of this trial.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Participants receive MUC1 peptide-poly-ICLC adjuvant vaccine subcutaneously (SC) in weeks 0, 2 and 10 and a booster injection in week 53.

ARM II: Participants receive saline SC in weeks 0, 2, and 10 and a booster injection in week 53.

After completion of treatment, patients are followed up every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* History of at least one of the following conditions in the previous 12 months:

  * Colorectal adenoma(s) >= 1 cm in maximal diameter
  * Colorectal adenoma(s) with villous or tubulovillous histology
  * Colorectal adenoma(s) with high grade (severe) dysplasia
* Presumptive evidence that all adenomatous lesions, including qualifying advanced adenoma, have been completely removed
* Ability to understand and the willingness to sign a written informed consent document
* Willingness to undergo screening tests and procedures
* Willingness to provide blood samples for toxicity monitoring and research purposes
* Not pregnant or nursing; note: a negative (serum or urine) pregnancy test must be documented =< 7 days prior to registration/randomization for women of childbearing potential
* Willingness to employ adequate contraception through week 53 of the study; note: women of childbearing potential and men must agree to use adequate contraception (hormonal, barrier method of birth control, abstinence) prior to study entry and for the period of active vaccination (through week 53); should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her physician immediately
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* Hemoglobin greater than 90% of the lower limit of institutional normal
* Platelets >= 100 B/L (10^9/L)
* White blood cell (WBC) > 2.5 B/L (10^9/L)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]), alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 x institutional upper limit of normal
* Alkaline phosphatase =< 1.5 x institutional upper limit of normal
* Total bilirubin =< 1.5 x institutional upper limit of normal
* Blood urea nitrogen (BUN) =< 1.5 x institutional upper limit of normal
* Creatinine =< 1.5 x institutional upper limit of normal
* Antinuclear antibody (ANA) test result excludes overt autoimmune disease; note: test result may be reported in any of the following formats: =< 1:160, negative, or < 1.0

Exclusion Criteria:

* History of any colorectal cancer
* History of other malignancy =< 5 years prior to the registration/randomization evaluation, with the exception of basal cell or squamous cell skin cancer
* Presence of an active acute or chronic infection or uncontrolled illness including, but not limited to unstable congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Acquired immunosuppressive diseases such as active human immunodeficiency virus (HIV) infection or congenital diseases of immunity
* History of heritable cancer syndrome (familial adenomatous polyposis [FAP], hereditary nonpolyposis colorectal cancer [HNPCC])
* History of auto-immune disease such as, but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, rheumatoid arthritis, ankylosing spondylitis, scleroderma, multiple sclerosis, Hashimoto's thyroiditis, or Grave's disease
* Current or planned use of immunomodulators including: infliximab, 6-MP (mercaptopurine), methotrexate, cyclosporine, or other immunomodulatory drugs
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the study agent
* Pregnant women
* Breastfeeding women
* Diagnosis of nonalcoholic steatohepatitis (NASH) and a NAFLD (nonalcoholic fatty liver disease) activity score (NAS) >= 5; NOTES and EXCEPTIONS: NAS is based on findings from a liver biopsy; participants with NAS of =< 2 are eligible for enrollment; participants with NAS of 3-4 must be discussed with the principal investigator and Division of Cancer Prevention (DCP) before enrollment to consider other risk factors (i.e., obesity, alcohol intake); participants with a prior diagnosis of NASH and no available NAS must be discussed with the principal investigator and DCP before enrollment to considered risk factors (i.e., obesity, alcohol intake)
* Receiving any other investigational agent =< 3 months prior to registration/randomization, except innocuous agents with no known interaction with the study agent (e.g., standard dose multivitamins or topical agents for limited skin conditions)
* Any use of oral corticosteroids =< 12 weeks prior to registration/randomization

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-06-23 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2026-03-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Schoen, Principal Investigator — Mayo Clinic
Locations (7):
- United States (6):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
- University of Puerto Rico, San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For the baseline discrepancy, we projected to enroll 120 patients originally, but only enrolled 110 in the end. Of the 110, only 102 completed the study and were evaluable for the primary endpoint. Of the 8 dropouts, 7 were cancels and 1 patient was a "withdrawal by subject".
Groups:
- Arm I (MUC1 Peptide-poly-ICLC Adjuvant Vaccine): Participants receive 300 microliters of MUC1 peptide vaccine SC in weeks 0, 2 and 10 and a booster injection in week 53.
- Arm II (Placebo): Participants receive identical-appearing placebo injection in weeks 0, 2, and 10 and a booster injection in week 53.
Period: Overall Study
Arm/Group | Arm I (MUC1 Peptide-poly-ICLC Adjuvant Vaccine) | Arm II (Placebo)
Started | 54 | 56
Received at Least One Dose of Treatment (Received at least one dose of treatment and assessed for AEs) | 53 | 50
Completed | 52 | 50
Not Completed | 2 | 6
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Cancel | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (MUC1 Peptide-poly-ICLC Adjuvant Vaccine) | Arm II (Placebo) | Total
Number analyzed (Participants) | 52 | 50 | 102
Age, Continuous [Median (Full Range); unit: years] | 59.5 [40.0 to 70.0] | 59.5 [47.0 to 70.0] | 59.5 [40.0 to 70.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 32 | 30 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 19
  Not Hispanic or Latino | 42 | 40 | 82
  Unknown or Not Reported | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 47 | 43 | 90
  Black or African American | 4 | 5 | 9
  Asian | 0 | 2 | 2
  Unknown: Patient unsure | 1 | 0 | 1
Performance status (PS) [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0) Fully active, able to carry on all pre-disease performance without restriction; 1) Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2) Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3) Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4) Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  Participants
    0 | 49 | 46 | 95
    1 | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Anti-MUC1 Immunoglobulin G (IgG) Levels as Determined by Enzyme-linked Immunosorbent Assay (ELISA)
Description: The ratio of the week 12 to week 0 IgG levels will be calculated and compared between the MUC1 vaccine and placebo. The Wilcoxon Rank-Sum test will be used. For all measurements of response (i.e. the primary endpoint), the 95% confidence intervals will also be provided.
Time Frame: Week 0 to week 12
Measure: Median (Full Range); unit: IgG ratio
Arm/Group | Arm I (MUC1 Peptide-poly-ICLC Adjuvant Vaccine) | Arm II (Placebo)
Number analyzed (Participants) | 52 | 50
IgG ratio | 1.2 [-0.5 to 17.3] | 1.0 [0.4 to 1.6]
Statistical Analysis 1: Comparison: Arm I (MUC1 Peptide-poly-ICLC Adjuvant Vaccine) vs Arm II (Placebo); Test type: Superiority; p = 0.0004, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Adenoma Recurrence Rate
Description: The secondary endpoint for Part 3 will evaluate the adenoma recurrence rate from surveillance exams. The rate is defined as the percentage of participants with adenoma recurrence.
Time Frame: At least one year and up to 3 years
Population: Participants who completed the surveillance exams were included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (MUC1 Peptide-poly-ICLC Adjuvant Vaccine) | Arm II (Placebo)
Number analyzed (Participants) | 48 | 47
percentage of participants | 56.3 | 66.0

3. Secondary Outcome: Booster Response
Description: The key secondary endpoint for Part 2 will assess the booster response at week 55 vs. week 52 for the vaccine as compared to placebo. The IgG ratios are summarized according to the following categories : <1, 1-<1.5, 1.5-<2, and >=2 (1-year response rate).
Time Frame: At week 55
Population: Participants with IgG levels at week 52 and 55 are included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MUC1 Peptide-poly-ICLC Adjuvant Vaccine) | Arm II (Placebo)
Number analyzed (Participants) | 51 | 44
Participants
  <1 | 17 | 18
  1- <1.5 | 15 | 22
  1.5- <2 | 2 | 2
  >=2 (1-Year Response Rate) | 17 | 2

4. Secondary Outcome: Participant-reported Injection Site Reactions - Redness at the Injection Site, Swelling/Induration, Itching at Site, and Skin Warmth at Site
Description: Participant-reported injection site reaction information is collected by the use of a participant-completed Vaccine Report Card. Participant-reported injection site reactions will be compared between study arms and are summarized below for redness at the injection site, swelling/induration, itching at site, and skin warmth at site.
Time Frame: Up to 55 weeks
Population: Participants who completed the Vaccine Report Card are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MUC1 Peptide-poly-ICLC Adjuvant Vaccine) | Arm II (Placebo)
Number analyzed (Participants) | 53 | 50
Participants
  Redness at the injection site: Yes | 36 | 2
  Redness at the injection site: None | 12 | 44
  Redness at the injection site: Missing | 5 | 4
  Swelling/induration: Yes | 30 | 0
  Swelling/induration: None | 18 | 46
  Swelling/induration: Missing | 5 | 4
  Itching at site: Yes | 17 | 1
  Itching at site: None | 31 | 45
  Itching at site: Missing | 5 | 4
  Skin warmth at site: Yes | 29 | 3
  Skin warmth at site: None | 19 | 43
  Skin warmth at site: Missing | 5 | 4

5. Secondary Outcome: Participant-reported Injection Site Reactions - Pain at the Injection Site Without Touching, and Tenderness (Pain at the Injection Site With Touch)
Description: Participant-reported injection site reaction information is collected by the use of a participant-completed Vaccine Report Card. Participant-reported injection site reactions will be compared between study arms and are summarized below for pain at the injection site without touching, and tenderness (pain at the injection site with touch).
Time Frame: Up to 55 weeks
Population: Participants who completed Vaccine Report Card are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MUC1 Peptide-poly-ICLC Adjuvant Vaccine) | Arm II (Placebo)
Number analyzed (Participants) | 53 | 50
Participants
  Pain at the injection site without touching: A lot | 1 | 0
  Pain at the injection site without touching: Some | 3 | 0
  Pain at the injection site without touching: A little | 33 | 0
  Pain at the injection site without touching: None | 16 | 50
  Tenderness (pain at the injection site with touch): A lot | 3 | 0
  Tenderness (pain at the injection site with touch): Some | 7 | 0
  Tenderness (pain at the injection site with touch): A little | 32 | 3
  Tenderness (pain at the injection site with touch): None | 11 | 47

6. Secondary Outcome: Number of Patients With at Least a 2-Fold Increase in the IgG Ratio
Description: The frequency and percentage of patients with at least a 2-fold increase in the IgG Ratio will be calculated and compared between the MUC1 vaccine and placebo. The Fisher's exact test will be used.
Time Frame: At 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (MUC1 Peptide-poly-ICLC Adjuvant Vaccine) | Arm II (Placebo)
Number analyzed (Participants) | 52 | 50
Participants | 13 | 0
Statistical Analysis 1: Comparison: Arm I (MUC1 Peptide-poly-ICLC Adjuvant Vaccine) vs Arm II (Placebo); Test type: Superiority; p = 0.0001, Fisher Exact

7. Other Pre Specified Outcome: Anti-MUC1 Antibody Titer by ELISA
Description: Comparisons between MUC1 and placebo will be performed using a two-sample t-test or Wilcoxon rank sum test, as appropriate. All categorical variables will be analyzed using chi-square tests or Fisher's exact test.
Time Frame: At approximately week 156
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Levels of Circulating MDSC in Peripheral Blood Mononuclear Cells by Flow Cytometry
Description: MDSC levels will be correlated with anti-MUC1 antibody levels and adenoma recurrence. Descriptive statistics and simple scatter plots will be generated to review the continuous biomarker data. In addition, for continuous biomarker values, the actual and percent change in the level of each of the biomarkers from baseline to post-baseline time points will be explored within each arm using Wilcoxon signed rank tests, and paired sample t-tests.
Time Frame: Baseline to up to 3 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in MUC1 Expression
Description: Descriptive statistics and simple scatter plots will be generated to review the continuous biomarker data. In addition, for continuous biomarker values, the actual and percent change in the level of each of the biomarkers from baseline to post-baseline time points will be explored within each arm using Wilcoxon signed rank tests, and paired sample t-tests.
Time Frame: Baseline to up to 3 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Establishment of a Biospecimen Repository Archive Including Live Cells, Plasma, and Germline DNA for Future Immunologic and Other Assays
Time Frame: Up to 3 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Incidence of Adverse Events as Graded by the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0.
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 3 years.
Description: All graded AEs are reported for patients who received at least 1 dose of treatment and assessed for AEs. Serious AE (SAE) reports may include any secondary serious or non-serious events considered related to the primary event (the reason for filing an expedited report); collectively, these events are referred to as Expedited AEs, and appear in the SAE table.
Arm/Group | Arm I (MUC1 Peptide-poly-ICLC Adjuvant Vaccine) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/50
Serious Adverse Events (participants affected / at risk) | 12/53 | 8/50
Other Adverse Events (participants affected / at risk) | 51/53 | 37/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (MUC1 Peptide-poly-ICLC Adjuvant Vaccine) (N=53) | Arm II (Placebo) (N=50)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 2 (2) | 1 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 1 (3)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 1 (1)
Renal calculi (Renal and urinary disorders) | 1 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (MUC1 Peptide-poly-ICLC Adjuvant Vaccine) (N=53) | Arm II (Placebo) (N=50)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 2 (2) | 0 (0)
Ear and labyrinth disorders - Oth spec (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (2) | 2 (3)
Eye disorders - Other, specify (Eye disorders) | 1 (2) | 0 (0)
Eyelid function disorder (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (5) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 5 (6) | 2 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (2)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Edema limbs (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 5 (7) | 3 (3)
Injection site reaction (General disorders) | 47 (150) | 10 (13)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) | 0 (0)
Autoimmune disorder (Immune system disorders) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 3 (3) | 2 (2)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 2 (2) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 4 (6) | 2 (3)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (4) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Cholesterol high (Investigations) | 2 (2) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1) | 2 (8)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 2 (2)
Joint range of motion decr cerv spine (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (5)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 2 (2)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Nystagmus (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Spasticity (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal calculi (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 1 (1)
Dyspareunia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Reproductive system and breast -Oth spec (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 7 (9) | 1 (4)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 2 (2) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 5 (5)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-22): https://cdn.clinicaltrials.gov/large-docs/25/NCT02134925/Prot_SAP_000.pdf